CLINICAL TRIAL: NCT06355375
Title: Exercise in Pregnancy and Risk of Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02.24
Record Dates: First submitted 2024-03-22; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Depression; Pregnancy Related
MeSH Terms: conditions — Depression | interventions — Exercise; Pregnancy

STUDY DESIGN:
Intervention Model Description: Exercise during pregnancy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Active Comparator): aerobic exercise during pregnancy
  Interventions: Behavioral: exercise in pregnancy
- no exercise (No Intervention): no recommendation regarding exercise

INTERVENTIONS:
Behavioral: exercise in pregnancy — aerobic exercise
  Arms: exercise

SUMMARY:
The prevalence of postpartum depression (PPD) varies between 11.9% and 19.2% during the perinatal period. PPD refers to minor and major depression incidents that occur during pregnancy or shortly after (up until 12 months after birth). The symptoms of PPD embrace feeling sad or having a depressed mood, being uninterested in the new-born, unreasonable crying and fear of injuring or harming the baby. Consequently, PPD can negatively impact the mother's well-being and the baby's development. The impact on a child can be short for cognitive and motor development . Although medication is a feasible alternative, many women have constraints due to continuing breastfeeding. Therefore, exercise can be an alternative that could help to deal with PPD. Exercise can be used as a preventive or treatment of mild depression at an early stage and as an addition to a treatment plan for major depressive disorder. Exercising during pregnancy and postpartum improves psychological health and also benefits physical fitness, weight gain control and the prevention or reduction of musculoskeletal discomfort and pain. Therefore, the American College of Obstetrics and Gynaecologists has recommended that women during pregnancy and postpartum engage in moderate-intensity physical activity almost every day for 30 min a day

DETAILED DESCRIPTION:
The prevalence of postpartum depression (PPD) varies between 11.9% and 19.2% during the perinatal period. PPD refers to minor and major depression incidents that occur during pregnancy or shortly after (up until 12 months after birth). The symptoms of PPD embrace feeling sad or having a depressed mood, being uninterested in the new-born, unreasonable crying and fear of injuring or harming the baby. Consequently, PPD can negatively impact the mother's well-being and the baby's development. The impact on a child can be short for cognitive and motor development . Although medication is a feasible alternative, many women have constraints due to continuing breastfeeding. Therefore, exercise can be an alternative that could help to deal with PPD. Exercise can be used as a preventive or treatment of mild depression at an early stage and as an addition to a treatment plan for major depressive disorder. Exercising during pregnancy and postpartum improves psychological health and also benefits physical fitness, weight gain control and the prevention or reduction of musculoskeletal discomfort and pain. Therefore, the American College of Obstetrics and Gynaecologists has recommended that women during pregnancy and postpartum engage in moderate-intensity physical activity almost every day for 30 min a day

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* low risk pregnancy
* age between 20 and 40

Exclusion Criteria:

* high risk pregnancy
* multiple gestation
* prior post partum depression
* any psychiatric disase
* controindication for exercise
* lung or heart disease
* prior preterm birth
* IVF pregnancy
* women who already perform agonistic sport activity

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 398 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
edinburgh depression scale | 3 months after delivery
  Edinburgh Postnatal Depression Scale (EDPS)

SECONDARY OUTCOMES:
Postpartum depression | 3 months after delivery
  DSM-5 (SCID-5)
preterm birth | 37 weeks of gestation
  defined as delivery before 37 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saccone G, Buonomo G, Ammendola A, Bardi L, Motta M, Gragnano E, Locci M. Exercise in Pregnancy and Risk of Postpartum Depression: A Randomised Controlled Trial. BJOG. 2026 Jan;133(2):211-217. doi: 10.1111/1471-0528.70010. Epub 2025 Sep 21. PMID 40976261